CLINICAL TRIAL: NCT05188235
Title: Pilot Study on the Evaluation of Sound Conduction of Healthy Infant Hips and Those With Developmental Dysplasia of the Hip (DDH)
Brief Title: Sound Conduction of Infant Hips
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study terminated upon departure of PI from Sponsoring Institution.
Sponsor: NYU Langone Health (Other)
Collaborators: University of Central Florida (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 21-01096
Record Dates: First submitted 2021-12-20; First posted 2022-01-12 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Developmental Dysplasia of the Hip
MeSH Terms: conditions — Developmental Dysplasia of the Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Infants with developmental dysplasia of the hip (Experimental): Infant participants putting on a device for 15 minutes to take different measurements of the hip
  Interventions: Device: Acoustical Resonance Device
- Infants without developmental dysplasia of the hip (Active Comparator): Infant participants putting on a device for 15 minutes to take different measurements of the hip
  Interventions: Device: Acoustical Resonance Device

INTERVENTIONS:
Device: Acoustical Resonance Device — Infants will be studied for 15 min using an electronic "tuning fork" to transmit sound through the hip from a point on the skin while transmitted sounds FDA-approved stethoscope

SUMMARY:
The objective of this study is to collect data that will be used to later design a method for the early diagnosis of diagnosis of developmental dysplasia of the hip (DDH).

DETAILED DESCRIPTION:
This will be a prospective study using an acoustic listening technique in combination with a standard clinical examination of DDH.

For both the clinical cases and healthy children that are enrolled, that all subjects will have an ultrasound completed for comparison to the use of the studied tuning fork method. The gold standard is POCUS (point of care ultrasound as performed by the pediatric orthopedic surgeon). Collected data will be compared to POCUS as performed by an expert and this is standard of care. Healthy subjects will be referred for evaluation and found to be healthy on subsequent US.

ELIGIBILITY:
Inclusion Criteria:

* Infants included in this study must be born at full term with a gestational age of 0-6 months
* Infants of both genders will be included
* Infants must have been screened for DDH.

Exclusion Criteria:

* Infants born prematurely
* Infants greater than six months of age.
* Nonviable neonates and neonates of uncertain viability

Ages: 1 Day to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 61 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2023-10-06 (Actual); Study Completion 2023-10-06 (Actual)

PRIMARY OUTCOMES:
Difference in soundwaves on the Actuator on patella, sensor on sacrum | Study visit 1 (Day 1)
  Descriptive statistics will be used to evaluate sound wave characteristics in infants with healthy hips. Inferential statistics will be used to compare the relationship between soundwave characteristics and diagnostic findings
Difference in soundwaves on the Actuator on patella, sensor on anterior superior iliac crest of pelvis | Study visit 1 (Day 1)
  Descriptive statistics will be used to evaluate sound wave characteristics in infants with healthy hips. Inferential statistics will be used to compare the relationship between soundwave characteristics and diagnostic findings
Difference in soundwaves on the Actuator on greater trochanter, sensor on sacrum | Study visit 1 (Day 1)
  Descriptive statistics will be used to evaluate sound wave characteristics in infants with healthy hips. Inferential statistics will be used to compare the relationship between soundwave characteristics and diagnostic findings
Difference in soundwaves on the Actuator on greater trochanter, sensor on anterior superior iliac crest | Study visit 1 (Day 1)
  Descriptive statistics will be used to evaluate sound wave characteristics in infants with healthy hips. Inferential statistics will be used to compare the relationship between soundwave characteristics and diagnostic findings

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Castaneda, MD, Principal Investigator — NYU Lagone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data.Upon reasonable request. Requests should be directed to study team members. To gain access, data requestors will need to sign a data access agreement.